CLINICAL TRIAL: NCT05244174
Title: Impact of Pancreatic Endoscopic Drainage on Exocrine Pancreatic Function in Patients With Unresectable Pancreatic Adenocarcinoma
Brief Title: Impact of Pancreatic Endoscopic Drainage on Exocrine Pancreatic Function in Unresectable Pancreatic Cancer
Acronym: DEPARA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, J. Enrique Domínguez-Muñoz, Director of Gastroenterology, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-006397-22
Record Dates: First submitted 2022-01-25; First posted 2022-02-17 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Neoplasm Malignant Head Primary; Pancreatic Exocrine Insufficiency
Keywords: pancreas cancer; ERCP; pancreatic exocrine insufficiency; pancreatic stent
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with pancreatic head adenocarcinoma will be randomized to biliary stent placement versus bilio-pancreatic stent placement using the computer-generated total randomization method. The randomization process will be carried out by one of the collaborating researchers who will not participate in the follow-up of patients
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One of the collaborator of the study will define which treatment group is assigned each patient (Group A and Group B). Only that investigator and the person who perform the ERCP (care provider) will know to which group is assigned the patient. Patients, investigators and outcome assessor are blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biliary stent (Active Comparator): Biliary stent by ERCP is indicated both in palliative treatment, because of biliary duct decompression improves patient comfort by decreasing itching and jaundice, as in the treatment of the disease itself, because of it lets reach non-toxic levels of bilirubin which is necessary for chemotherapeutic treatment.
  Interventions: Device: Pancreatic stent
- Biliary and pancreatic stent (Experimental): During ERCP, the cannulation of the main pancreatic duct may be performed for the placement of a pancreatic duct stent, which is performed routinely as a prophylaxis of post-ERCP acute pancreatitis in patients at risk. In patients with pancreatic cancer, the placement of a pancreatic stent could improve pancreatic secretion by clearing the main pancreatic duct and thus it could improve fat digestion and nutritional status of patients, avoiding the need for PERT
  Interventions: Device: Pancreatic stent

INTERVENTIONS:
Device: Pancreatic stent — Insertion of a pancreatic stent during ERCP to improve pancreatic secretion

SUMMARY:
Background: exocrine pancreatic insufficiency (IPE), frequent in patients with pancreatic cancer, plays a major role in malnutrition and cachexia with a significant impact on survival, quality of life and tumor progression. IPE due to obstruction of the main pancreatic duct and atrophy of pancreatic parenchyma proximal to the tumor could be corrected by insertion of a pancreatic stent for improving nutritional status and consequently survival.

Aim: The aim of this study is to assess the impact of transpapilar drainage of the main pancreatic duct on exocrine pancreatic function, nutritional status, and life survival in patients with unresectable pancreatic adenocarcinoma.

Methods: Impact of pancreatic endoscopic drainage on exocrine pancreatic function in patients with unresectable pancreatic adenocarcinoma (DEPARA) is a double-blind, prospective, multicentre, international clinical trial. Unresectable locally advanced or metastatic pancreatic cancer (PDAC) will be diagnosed according to the National Comprehensive Cancer Network (NCCN) criteria and the indication of endoscopic retrograde cholangiopancreatography (ERCP) due to obstructive jaundice (>3mg/dl). PEI will be defined by reduced fecal elastase levels. The nutritional status will be determined by means of Mini-Nutritional Assessment score, sarcopenia score (SARC-F) and laboratory blood tests. Primary aim: Evaluation of the improvement and difference of pancreatic secretion as measured by fecal elastase at 2 weeks post-stenting (biliopancreatic versus biliary). Secondary aims: evaluation of the prevalence of PEI post-stenting (biliopancreatic versus biliary) and proportion of patients normalizing pancreatic function. The difference in terms of weight loss, maldigestion symptoms, GI-Qol, nutricional status and performance status. Survival at 2 weeks, 3 and 6 months, overall survival. Analyzes: fecal elastase value at 2 weeks post-stenting (absolute value of fecal elastase) compared between biliopancreatic stent group and biliary stent group.

Discussion: DEPARA will provide insight into the role of pancreatic stents for PEI, malnutrition and progression-free survival in the outcomes of PDAC unresectable.

DETAILED DESCRIPTION:
In a recent study by our group, 13 patients with unresectable pancreatic head cancer and PEI were randomized into 2 groups (biliopancreatic stent versus biliary stent), showing a statistically significant improvement in exocrine pancreatic function in favor of biliopancreatic drainage (absolute increase 13C-CRR 23.75% (CI 9.62, 31.74%) vs -1.92% (CI -4.17, 13.92%) p=0.015). All patients who underwent pancreatic drainage showed normalization of pancreatic function and nutritional parameters.

A randomized clinical trial is being conducted in patients with unresecable pancreatic cancer to evaluate the effectiveness of pancreatic stent placement in improving pancreatic secretion by desobstructing the main pancreatic duct and thus improving digestion, nutritional status and consequently patient survival.

HYPOTHESIS:

Transpapillary pancreatic drainage with a pancreatic stent is associated with a significant improvement in pancreatic function, nutritional status, maldigestion symptoms and quality of life in patients with unresectable pancreatic adenocarcinoma who require endoscopic bile duct drainage.

AIM:

To investigate the impact of transpapillary drainage of the pancreatic duct on exocrine pancreatic function, nutritional status, maldigestion symptoms and quality of life in patients with unresectable pancreatic adenocarcinoma.

METHODS:

Patients diagnosed with unresectable pancreatic adenocarcinoma according to the NCCN criteria that have an indication of performing an endoscopic retrograde cholangiopancreatography (ERCP) due to the presence of obstructive jaundice (>3mg/dL).

VARIABLES:

The following variables will be recorded in a dedicated Case Report Form (CRF). All these measures are part of a standard workup of advanced PDAC patients and considered good clinical practice.

• Patient-related: Sex, race, age at diagnosis Significant comorbilities: chronic kidney failure, chronic heart failure, or respiratory insufficiency requiring oxygen treatment

Mini-Nutritional Assessment (MNA) score. Primarily developed for elderly patients, MNA score was successfully used in the PreMiO study (Prevalence of malnutrition in patients at first medical oncology visit) to identify the risk of malnutrition or malnutrition among cancer patients at their first medical oncology visit:

1. 0-7 points: Malnourished
2. 8-11 points: At risk of malnutrition
3. 12-14 points: Normal nutritional status Sarcopenia score (SARC-F score) Cachexia [weightloss >5% in the las 6 months or weightloss >2% if IMC<20kg/m2] 12-item functional assessment of anorexia/cachexia therapy anorexia/cachexia subscale (FAACT-A/CS-12) Performance Status-ECOG European Organization for Research and Treatment of Cancer (EORTC) QLQ-PAN26 scale (22) A biliary, duodenal or pancreatic stent Date of diagnosis, visit 1, visit 2 (2 weeks), visit 3(3 months), visit 4 (6 months) and death/loss from follow-up .

   Check up on survival at third month and sixth month Chemotherapy regimen

   • Tumor-related: Tumor site documented by endoscopic ultrasound, CT, or magnetic resonance imaging (head, body, or tail) Stage according to National Comprehensive Cancer Network (NCCN) criteria

   • Nutritional parameters: C-reactive protein, total protein, albumin, cholesterol, iron, transferrin, ferritin, magnesium, zinc Blood fasting glucose, glycated hemoglobin

   • Pancreatic function and treatment: PEI will be defined by levels of fecal elastase-1 <200 mcg/g; pancreatic enzyme replacement therapy (PERT), date of starting PERT, the dosage of daily taken PERT Diabetes mellitus (DM), date of DM diagnosis, DM type, DM treatment

   • Therapy-related (endoscopic procedure): ERCP will be performed under deep sedation by expert endoscopists. Endoscopic biliary sphincterotomy will be performed in all cases before biliary drainage. Partially or fully covered self-expandable metal biliary stents of 10mm in diameter (Wallstent RX biliary Stent System, Boston Scientific, Marlborough, Massachusetts, USA) will be used. Stent length will be selected to cover the length of the biliary stenosis. In patients allocated to pancreatic drainage, plastic pancreatic 7 to 10Fr straight stents (AdvanixTMand NaviFlexTM RX Pancreatic Delivery System, Boston Scientific, Marlborough, Massachusetts, USA) will be used. Stent length will be selected to cover the length of the pancreatic stenosis. Pancreatic sphincterotomy will be performed before pancreatic drainage if required.

   STUDY PERIOD Depending on approval of the Local Ethics Committees, enrollment is planned to start from Februrary 2023 and last until November 2023 or until the planned power calculation has been met.

   DESCRIPTION OF THE INTERVENTION (SCHEDULE OF VISITS) Patients with pancreatic head adenocarcinoma will be randomized to biliary stent placement versus bilio-pancreatic stent placement using the computer-generated total randomization method. The randomization process will be carried out by one of the collaborating researchers who will not participate in the follow-up of patients Screening visit (Hospitalization Unit) After diagnosis of locally advanced or metastatic pancreatic head adenocarcinoma, the investigator in charge of the study will evaluate the inclusion and exclusion criteria and will give the explanation of the study to the patients and delivery of informed consent.

   Visit 1 (inclusion and exclusion criteria evaluation, IC signature, baseline data collection)

   After the signature of the consent and the collection of the baseline data, all patients will do a complete analysis with nutritional parameters and FE-1 test. Nutritional scores and quality of life scores will be evaluated. Then, they will be randomized into the bilio-pancreatic stent group or biliary stent group. Patients randomized to the first group in which pancreatic cannulation is not achieved will be included in the biliary stent group in the protocol analysis. Patients in whom biliary cannulation is failed will be excluded because they need other techniques for biliary drainage.

   Visit 2 (2 weeks after ERCP) A new determination of FE-1 will be made. In patients with a fecal concentration of elastase<100 µg/g, substitutive enzymatic treatment will be administered according to clinical guidelines and standard clinical practice (70,000 U.Ph. with main meals and 35,000 U.Ph. with minor meals).

   Visit 3 (3 months after ERCP) A new analysis will be made with nutritional parameters. Nutritional scores and quality of life scales will be analyzed.

   Visit 4 (6 months after ERCP) A new analysis will be made with nutritional parameters. Again, nutritional and quality of life scales will be evaluated MEDICATION OF THE STUDY The use of pancreatic enzyme replacement treatment will be recorded as well as data regarding the employed chemotherapy regimen.

   STATISTICAL ANALYSIS The data will be represented in absolute number or percentage, with their respective mean and standard deviation, median and interquartile range as a function of their distribution.

   Qualitative variables will be compared between both groups by chisquare test or Fisher's exact test as appropriate.

   Continuous variables will be compared using a Mann Whitney U test for independent samples.

   A logistic regression model will be created to know which factors are independently associated with the development of IPE (tumor size, tumor stage, main pancreatic duct dilation, pancreatic parenchymal atrophy).

   A proportional risk analysis of Cox will be performed to compare survival in both treatment groups.

   A value of <0.05 will be considered statistically significant All data will be anonymous once data collection is completed, respecting the confidentiality of the subjects participating, in accordance with data protection laws. All analyses will be performed in STATA 16 (Statacorp LLC, Texas).

   POWER SIZE CALCULATION Based on data from our pilot study that included 20 patients with unresectable pancreatic head adenocarcinoma in which a difference in the FE-1 test of 96mcg/g (SD=151) between the two treatment groups was showed. Assuming an alpha error=0.05 and 80% potency, it would be necessary to include 39 patients in each treatment group. Given the nature of the pathology there is the possibility of a 5% loss, so the total estimated sample size would be 82 patients.

   DISCUSSION Given the sparse overall scientific data on the subject, the investigators have designed a clinical trial that addresses the impact of pancreatic stent on pancreatic secretion, nutritional status and survival of patients with advanced PDAC unresectable. DEPARA will be the first targeted study for investigating whether pancreatic stents positively influence nutritional status and survival of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological diagnosis of PDAC
* Radiological diagnosis of the advanced stage not suitable for upfront surgical resection (either locally advanced or metastatic)
* Endoscopic biliary drainage required due to obstructive jaundice
* A written consent to participate in the study

Exclusion Criteria:

* Known history of chronic pancreatitis
* Any contraindication for ERCP under deep sedation or impossibility of biliary cannulation.
* Inclusion in a clinical trial 4 weeks before this study.
* Poor performance status (Eastern Cooperative Oncology Group scale (ECOG) =4)
* Known history of gastrointestinal or pancreatic surgery that is associated with alteration of -pancreatic function.
* Known history of chronic bowel disease (inflammatory bowel disease) that could be associated with nutrient malabsorption
* Gastrointestinal obstruction caused by tumor.
* Pregnancy or breastfeeding
* Unwillingness or inability to understand the study and sign the consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Level of Fecal elastase-1 | 1 month after ERCP
  Evaluation of the efficacy of the endoscopic insertion of biliopancreatic stent compared to biliary stent in the improvement of pancreatic secretion measured by FE-1 test in patients with unresectable pancreatic cancer

SECONDARY OUTCOMES:
Quality of life (QoL) | At 3 and 6 months after ERCP
  Quality of life and differences between both groups. It will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-PAN26 scale. Minimun of the scale 25 points, maximum 100. Higher puntuations are related to worse outcome.
Nutritional status | At 3 and 6 months after ERCP
  Nutritional status in each treatment group using the Patient-Generated-Subjective Global Assessment (PS-GHS). Minimum of the scale 0 points. Maximum >9 points. Higher puntuations are related to worse outcome
Body weight | At 3 and 6 months after ERCP
  Difference in body weight between each of the treatment groups
Survival | At 6 months
  Survival of patients with unresectable pancreatic adenocarcinoma in the group with biliopancreatic stent vs biliary stent.
Prevalence of PEI | 1 month, 3 and 6 months
  Prevalence of PEI post-stenting measured by fecal elastase.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Dominguez Munoz, MD, Principal Investigator — University Hospital of Santiago de Compostela
Locations (1):
- Daniel de la Iglesia, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No